CLINICAL TRIAL: NCT05146661
Title: An In-hospital Feasibility Study of the NEURESCUE Device as an Adjunct to Cardiac Arrest
Brief Title: NEURESCUE Device as an Adjunct to Cardiac Arrest
Acronym: ARISE-EU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: neurescue (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Safestudy5
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest; Cardiovascular Diseases
MeSH Terms: conditions — Heart Arrest; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The NEURESCUE device will be used as an adjunct to ALS.
  Interventions: Device: NEURESCUE device

INTERVENTIONS:
Device: NEURESCUE device — The balloon catheter is delivered via the femoral artery, temporarily inflating a soft balloon in the descending to redirect blood flow towards the upper body.

SUMMARY:
The NEURESCUE device is the first intelligent balloon catheter for aortic occlusion, an emergency technique that supercharges blood flow to the heart and brain within one minute from deployment.

The catheter-based device is delivered via the femoral artery, temporarily inflating a soft balloon in the descending to redirect blood flow towards the upper body.

The objective of the study is to investigate the safety and performance of the NEURESCUE device as an adjunct to Advanced Life Support (ALS) in adults with cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤79 years
2. Witnessed cardiac arrest
3. CPR initiated within 7 min of presumed arrest
4. Cardiac arrest not responding to standard ALS
5. Total CPR time ≤ 40 min at the time of screening for enrollment

Exclusion Criteria:

1. Traumatic cardiac arrest
2. Known pregnancy
3. Known terminal disease
4. Known Do-Not-Resuscitate (DNR) order
5. Subjects whose femoral arterial access site cannot accommodate an 8 Fr introducer sheath
6. Subjects currently on mechanical circulatory support

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Successful balloon inflation within 10 minutes from first vessel puncture | Assessed up to 10 min

SECONDARY OUTCOMES:
Change in central blood pressure | At the initiation of balloon inflation compared to two minutes after finalizing balloon inflation
Total cardiopulmonary resuscitation (CPR) time at the screening for enrollment | From initiation of cardiopulmonary resuscitation (CPR) to screening for enrollment
Total ALS time at initiation of the investigational procedure | From initiation of ALS to initiation of the investigational procedure
Time from first vessel puncture to successful sheath insertion | From first needle stick to successful sheath insertion
Rate of occlusion success | Assessed up to 1 hour
Return of spontaneous circulation (ROSC) | Assessed up to 1 hour
  The endpoint is dichotomous (yes/no) for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Michael Preusch, M.D., Principal Investigator — University Hospital Heidelberg
Locations (2):
- Germany (2):
  - Charité - Universitätsklinikum Berlin, Berlin
  - Universitätsklinikum Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: No
Individual request